CLINICAL TRIAL: NCT05475821
Title: A First in Human, Single Ascending Dose Study for the Assessment of Pharmacokinetics, Safety and Tolerability of ABBV-990 in Healthy Male and Female Subjects
Brief Title: Study to Assess Adverse Events and How Oral ABBV-990 Moves Through the Body of Adult Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision: re-evaluation of risk vs benefit (based on animal data)
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: M23-661
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CoronaVirus Disease-2019 (COVID-19); ABBV-990; SARS-CoV-2; Severe Acute Respiratory Syndrome Coronavirus-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Group 1 (Experimental): Participants will receive ABBV-990 Dose A or matching placebo.
  Interventions: Drug: ABBV-990; Drug: Placebo for ABBV-990
- Group 2 (Experimental): Participants will receive ABBV-990 Dose B or matching placebo.
  Interventions: Drug: ABBV-990; Drug: Placebo for ABBV-990
- Group 3 (Experimental): Participants will receive ABBV-990 Dose C or matching placebo.
  Interventions: Drug: ABBV-990; Drug: Placebo for ABBV-990
- Group 4 (Experimental): Participants will receive ABBV-990 Dose D or matching placebo.
  Interventions: Drug: ABBV-990; Drug: Placebo for ABBV-990
- Group 5 (Experimental): Participants will receive ABBV-990 Dose E or matching placebo.
  Interventions: Drug: ABBV-990; Drug: Placebo for ABBV-990

INTERVENTIONS:
Drug: ABBV-990 — Oral Tablet
Drug: Placebo for ABBV-990 — Oral Tablet

SUMMARY:
This study will assess how safe ABBV-990 is and how ABBV-990 moves through the body of adult healthy participants. Adverse Events will be assessed.

ABBV-990 is an investigational drug being developed for the treatment of SARS-CoV-2 infections. Participants are randomly assigned to one of the 5 treatment groups. Each group receives different treatment. There is 1 in 4 chance that participants are assigned to placebo. Approximately 40 adult healthy volunteers will be enrolled in a single site in the United States.

Participants will receive oral tablet of ABBV-990 or matching placebo on Day 1 and followed for approximately 30 days.

Participants will be confined for 5 days. Adverse Events and blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) is >= 18.0 to <= 32.0 kg/m2.
* Laboratory values meet the protocol-specified criteria.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG).
* In the opinion of the investigator, participant is a suitable candidate for enrollment in the study.

Exclusion Criteria:

* Have any clinically significant ECG abnormalities.
* History of any clinically significant sensitivity or allergy to any medication or food.
* Known active SARS-CoV-2 infection at screening and upon initial confinement.
* History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.
* Currently enrolled in another interventional clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 30 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.
Maximum Observed Plasma Concentration (Cmax) of ABBV-990 | Up to approximately 5 days
  Cmax of ABBV-990.
Time to Cmax (Tmax) of ABBV-990 | Up to approximately 5 days
  Tmax of ABBV-990.
Apparent Terminal Phase Elimination Rate Constant (β) of ABBV-990 | Up to approximately 5 days
  Apparent terminal phase elimination rate constant of ABBV-990.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-990 | Up to approximately 5 days
  Terminal phase elimination half-life of ABBV-990.
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Time of the Last Measurable Concentration (AUCt) of ABBV-990 | Up to approximately 5 days
  AUCt of ABBV-990.
AUC From Time 0 to Infinite Time (AUCinf) of ABBV-990 | Up to approximately 5 days
  AUCinf of ABBV-990.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 247995, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-661